CLINICAL TRIAL: NCT03257930
Title: Percutaneous Ethanol Injection for Benign Cystic Thyroid Nodules
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: hassan harby mohamed (Other)
Responsible Party: Sponsor-Investigator, hassan harby mohamed, general surgery, Assiut University
Organization: Assiut University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Ethanol Injection
Record Dates: First submitted 2017-08-17; First posted 2017-08-22 (Actual); Last update posted 2020-05-15 (Actual); Status verified 2020-05

CONDITIONS: Thyroid Nodule
MeSH Terms: conditions — Thyroid Nodule | interventions — Ethanol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- injection of ethanol (Experimental): use of ethanol injection in the treatment of cystic thyroid nodule
  Interventions: Drug: ethanol injection

INTERVENTIONS:
Drug: ethanol injection — inject ethanol in cystic thyroid nodule and follow up until complete recovery

SUMMARY:
Use of ethanol injection in treatment of cystic thyroid nodule

DETAILED DESCRIPTION:
Thyroid nodules are common discreet lesions in the parenchyma of thyroid gland which can either be palpated or made out during imaging like ultrasonography (USG).Clinically palpable thyroid nodules have a prevalence of 4-7% in the general population . However, the prevalence increases to 20-76% when USG is used for detection.

Goiter and the associated thyroid nodules result in anxiety, cosmetic disfigurement, and rarely compressive symptoms necessitating surgical removal, a procedure inherently associated with risks and complications Percutaneous sclerotherapy has been suggested to be an effective alternative, especially in patients with cystic nodules. Simple cystic (purely cystic) constitutes 6-28% of all thyroid nodules, are usually benign, filled with cellular debris or blood, and are a result of degeneration or hemorrhage into a hyperplastic nodule.

Among the various compounds (sodium tetradocyl sulfate, hydroxypolyethoxydodecan, tetracycline, and ethanol) tried for sclerosis of cystic thyroid nodules, outcomes are best and most studied with ethanol. However, data on outcomes of percutaneous aspiration and ethanol injection (PEI) in resolution of thyroid nodules is highly variable in different studies (success rate: 38-85%), which may be due to different populations studied and the heterogeneous nature of thyroid nodules evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. Adult male or female patient with cystic thyroid nodule
2. Presence of pressure symptoms or cosmetic problems
3. Benign lesions confirmed by histopathological examination by FNAC.
4. Serum levels of thyroid hormone thyrotropin, within normal limits.

Exclusion Criteria:

1. Nodules showing malignant features(ie, speculated margin, markedly hypo echoic, micro- or macro calcifications) at US
2. solid thyroid nodule
3. mixed thyroid nodule(cystic with solid component)

Ages: 15 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 1 (Actual)
Dates: Start 2017-08-11 (Actual); Primary Completion 2018-07-11 (Actual); Study Completion 2019-01-01 (Actual)

PRIMARY OUTCOMES:
Reduction of volume of the cyst about 96.9% | Reduction of volume of the cyst about 96.9% within 6 month
  Reduction of volume of the cyst about 96.9%

SECONDARY OUTCOMES:
symptomatic improvement | 3 month
  cosmetic improvement of the ugly appearance of the cyst from the neck

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut University, Asyut, Egypt

REFERENCES:
- [Background] Vogel D, Durham AC, de Marcillac GD. Metastable aggregates in the polymerisation of tobacco-mosaic-virus protein. Eur J Biochem. 1977 Sep 15;79(1):161-71. doi: 10.1111/j.1432-1033.1977.tb11794.x. No abstract available. PMID 21087
- [Background] Monzani F, Lippi F, Goletti O, Del Guerra P, Caraccio N, Lippolis PV, Baschieri L, Pinchera A. Percutaneous aspiration and ethanol sclerotherapy for thyroid cysts. J Clin Endocrinol Metab. 1994 Mar;78(3):800-2. doi: 10.1210/jcem.78.3.8126160.